CLINICAL TRIAL: NCT06390787
Title: Enhancing Antiemetic Efficacy: A Randomized Trial of Vitamin B6 and Metoclopramide Combination Therapy Versus Traditional Regimens
Brief Title: The Efficacy of B6 and Metoclopramide Combination in Comparison With the Other Antiemetics
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2024-04-21; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Vomiting
Keywords: Vomiting; B6 Vitamin; Metoclopramide; Zofran
MeSH Terms: conditions — Vomiting | interventions — Metoclopramide; Vitamin B 6; Pyridoxine; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Metoclopramide Group (Active Comparator): This group of 50 patients with vomiting were given Metoclopramide only for vomiting.
  Interventions: Drug: Metoclopramide
- Zofran Group (Active Comparator): This group of 50 patients with vomiting were given Zofran only for vomiting.
  Interventions: Drug: Ondansetron
- B6 and Metoclopramide Group (Experimental): This group of 50 patients with vomiting were given B6 and Metoclopramide combination for vomiting.
  Interventions: Drug: Metoclopramide and Vitamin B6
- Control Group (No Intervention): This group of 50 patients with vomiting were given nothing for vomiting.
- Vitamin B6 Group (Active Comparator): This group of 50 patients with vomiting were given Vitamin B6 only for vomiting.
  Interventions: Drug: Vitamin B6

INTERVENTIONS:
Drug: Metoclopramide and Vitamin B6 — We gave a combination of vitamin B6 (pyridoxine) and metoclopramide as a treatment for managing nausea and vomiting.
  Other Names: Vitamin B6 and Metoclopramide combination
  Arms: B6 and Metoclopramide Group
Drug: Vitamin B6 — We gave only vitamin B6 (pyridoxine) as a treatment for managing nausea and vomiting.
  Other Names: Pyridoxine
  Arms: Vitamin B6 Group
Drug: Ondansetron — We gave only Zofran as a treatment for managing nausea and vomiting.
  Other Names: Zofran
  Arms: Zofran Group
Drug: Metoclopramide — We gave only Metoclopramide as a treatment for managing nausea and vomiting.
  Other Names: Plasil
  Arms: Metoclopramide Group

SUMMARY:
This study investigates the effectiveness of combining vitamin B6 (pyridoxine) and metoclopramide compared to standard antiemetic treatments for managing nausea and vomiting. Through a prospective, randomized controlled trial involving adult patients with diverse causes of nausea and vomiting, we aim to evaluate the frequency, severity, and tolerability of the B6 and metoclopramide combination. By elucidating its comparative efficacy against established antiemetics, this research seeks to provide evidence-based guidance for clinicians in selecting optimal treatment regimens tailored to individual patient needs, ultimately enhancing the management of nausea and vomiting across various medical conditions.

DETAILED DESCRIPTION:
Title: Investigating the Efficacy of B6 and Metoclopramide Combination Versus Alternative Antiemetics: A Clinical Trial Proposal

Introduction:

Nausea and vomiting are common symptoms across various medical conditions and can significantly impact patients' quality of life and treatment outcomes. While several antiemetic medications exist, finding the most effective regimen remains a clinical challenge. This proposal aims to investigate the efficacy of a combination therapy comprising vitamin B6 (pyridoxine) and metoclopramide compared to other antiemetics in managing nausea and vomiting.

Rationale:

Both vitamin B6 and metoclopramide have shown antiemetic properties through different mechanisms of action. However, the comparative efficacy of this combination therapy against other standard antiemetics remains largely unexplored. Understanding the relative effectiveness of this combination could provide valuable insights into optimizing antiemetic strategies, particularly in patients with chemotherapy-induced nausea and vomiting (CINV), postoperative nausea and vomiting (PONV), and other related conditions.

Objectives:

This prospective, randomized controlled trial aims to evaluate the efficacy of B6 and metoclopramide combination therapy compared to alternative antiemetic regimens in reducing the frequency and severity of nausea and vomiting episodes in adult patients. Additionally, the study seeks to assess the safety profile and tolerability of the combination therapy.

Conclusion:

By elucidating the comparative efficacy of B6 and metoclopramide combination therapy, this study endeavors to contribute to evidence-based decision-making in the management of nausea and vomiting. The findings could potentially guide clinicians in selecting the most appropriate antiemetic regimen tailored to individual patient needs, ultimately improving patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Any patients with vomiting

Exclusion Criteria:

* Patients vitally unstable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
Nausea | 1 day
  Four characteristics of nausea typically were measured including duration, frequency, severity, and associated distress. Duration was measured by asking the patient if they had experienced nausea and/or the number of hours that nausea was experienced during the time frame addressed.
Vomiting | 1 day
  Four characteristics of vomiting typically were measured including duration, frequency, severity, and associated distress. Duration was measured by asking the patient if they had experienced vomiting and/or the number of hours that vomiing was experienced during the time frame addressed.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Talib T Hashim, MBChB, Principal Investigator — University of Warith Al-Anbiyaa, College of Medicine
Locations (1):
- Al-Nassiryah Teaching Hospital, Nasiriyah, Thi Qar, Iraq

IPD SHARING:
Plan to Share IPD: No
We are not sharing any individual data with anyone.